CLINICAL TRIAL: NCT03876600
Title: Cost-utility Analysis of Ambulatory Care Compared to Conventional Patient Care of Permanent Pacemakers Replacement for Elective Replacement Indicator
Acronym: START
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nantes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RC18_0034
Record Dates: First submitted 2019-02-14; First posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Pacemaker Ddd
Keywords: pacemaker; replace for elective wear; french context; cost-utility analysis; prospective; multicentric; randomized study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional hospitalization management. (Experimental): The patients who are randomized to have a conventional hospitalization for the pacemaker replacement have conventional management.
  In this management patient come to hospital one day before this surgical operation and he is operated next day
  Interventions: Procedure: Replacement of permanent pacemakers for elective wear.
- ambulatory management (Active Comparator): The patients who are randomized to have a ambulatory surgery for the pacemaker replacement have ambulatory management.
  In the ambulatory hospitalization patients come to hospital and have a surgical operation the same day
  Interventions: Procedure: Replacement of permanent pacemakers for elective wear.

INTERVENTIONS:
Procedure: Replacement of permanent pacemakers for elective wear. — START's intervention is a replacement of permanent pacemakers for elective wear, for the both arms the surgical intervention is the same. The surgical procedure is the same in the both arms.
  The differences are in conventional hospitalization, patient comes to hospital one day before operation and he can go out one day after operation. In ambulatory patient come to hospital operation days and he can got out the same day.

SUMMARY:
START study is a comparison of cost-utility between permanent pacemaker replacement ambulatory care and permanent pacemaker replacement conventional hospitalization care.

The hypothesis of the study is that ambulatory care compared to conventional hospitalization, involving a stay of more than 24 hours, would reduce hospitalization and care expenses without loss of quality of care and without increasing the complication rate for patients.

DETAILED DESCRIPTION:
In France, nearly 49,000 permanent pacemakers are implanted each year. The pacemaker longevity is about 10 years which leads to their replacement.

In France, in 2016, 15,764 pacemaker replacement hospital stays took place. 10.6% of them were made during an outpatient stay, 12.4% during a one-night hospitalization and 70.7% during hospitalization for two or more than two nights for the severity level 1.

If the outpatient care management is deployed at 90%, the economy of the cost care will be estimated to be 3,5 million euros and a reduction of 15 582 hospitalization night's stay.

The aim of START study is to compare cost-utility between ambulatory and conventional hospitalization care of permanent pacemakers replacement for elective replacement indicator and to demonstrate equivalence between outpatient management and conventional hospitalization management.

This study is in adequation with the national ambition to deploy the outpatient management in France. Surgery is the same with both hospitalization managements.

An ambulatory surgery need to present different advantages and benefits like high quality care and substantial cost savings.

The benefits of ambulatory care management are :

* An economy of hospitalization nights cost.
* A decrease in health costs related to the surgery realization.
* Patient satisfaction expected due to hospital discharged within 24 hours. Patient is expected to go home the same day as the surgery with good perception of ambulatory surgery.
* A decrease in the disorientation risk in the elderly patient is also expected.

Surgery is the same with both hospitalization managements.

Patients will be randomized in 2 arms. An arm conventional hospitalization management (control arm) and an arm outpatient care management.

Study period is 30 months. Patients will be following during 6 months. The recruitment time will be 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over 18 years old.
* Replacement of permanent pacemakers for battery elective wear without programmed act in the sensors regardless of pacemaker type, simple, dual or triple chambers and regardless pacemaker label.
* Patient living less than an hour from a hospital center
* Patient is able to answer the phone.
* Patient has an accompaniment the go out night
* Pacemaker-dependent patient or not regardless of indication of placement of the pacemaker
* Patient with or without anticoagulant treatment: the anticoagulant treatment is managed by center under these habits.
* Patient has given this free and informed consent.
* Patient having insurance in France.

Exclusion Criteria:

* Ambulatory Hospitalization is impossible.
* Patient refuses to participate
* Patient has hemostasis disorder yielding ambulatory hospitalization impossible.
* Woman is pregnant, nursing mothers or the patient don't receive an effective contraception.
* Patient under guardianship, safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Cost-utility analysis,from the perspective of the society and a time horizon of 6 months,of ambulatory management compared to the intervention in conventional hospitalization of a replacement,for elective wear,permanent pacemakers | 6 month
  Incremental cost-utility ratio (cost by quality-adjusted life-years, QALY) of outpatient management compared to compared to the intervention in conventional hospitalization (≥1 night) of a replacement, for elective wear, permanent pacemakers. This analysis is from the perspective of the society and a time horizon of 6 months.

SECONDARY OUTCOMES:
Assess, the point of view of health insurance and health care institutions with a time horizon of 5 years, the annual and global budgetary impact in € of different diffusion scenarios for ambulatory to replace conventional hospitalization | on a time horizon of 5 years
  Annual and global net profit cost in € of different diffusion scenarios for ambulatory to replace conventional hospitalization.
Evaluate and compare the rate of complications of different management within 6 months after the intervention in both arms. | on time horizon of 6 months
  Complication statement requiring a rehospitalization with reoperation. This objective is assessed by the complication statement requiring rehospitalization without reoperation and complication with not requiring rehospitalization.
Evaluate the ambulatory failure rate | during all the study, during 30 months.
  Ambulatory failure rate. It is a ratio of the number of ambulatory visits converted to conventional hospitalization and the total number of ambulatory visits.
Evaluate and compare patients satisfaction between intervention and hospital management in both arms | during hospitalization, during 2 days
  Satisfaction with the intervention and management at the hospital with questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Probst, Principal Investigator — Nantes University Hospital
Locations (14):
- France (14):
  - Lyon University Hospital, Lyon, Bron
  - Angers University Hospital, Angers
  - Brest University Hospital, Brest
  - Dijon University Hospital, Dijon
  - Grenoble University Hospital, Grenoble
  - AP-HM, Marseille
  - Montpellier University Hospital, Montpellier
  - Nancy University Hospital, Nancy
  - AP-HP, La Pitié Salpétrière, Paris
  - Rennes University Hospital, Rennes
  - Saint-Etienne University Hospital, Saint-Etienne
  - Strasbourg University Hospital, Strasbourg
  - Toulouse University Hospital, Toulouse
  - Tours University Hopsital, Tours

IPD SHARING:
Plan to Share IPD: No